CLINICAL TRIAL: NCT03006081
Title: The Efficacy of Intravitreal Aflibercept Injection in Improvement of Retinal Nonperfusion in Patients With Diabetic Retinopathy
Brief Title: The Efficacy of Intravitreal Aflibercept Injection in Improvement of Retinal Nonperfusion in Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young Hee Yoon, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLOW_001
Record Dates: First submitted 2016-12-05; First posted 2016-12-30 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2018-12

CONDITIONS: Diabetic Retinopathy
Keywords: Retinal nonperfusion; Aflibercept
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2mg intravitreal aflibercept injection (Experimental): 2mg intravitreal aflibercept (Eylea) injection at baseline, 1M, 2M, 3M, 4M, and 5M
  Interventions: Drug: Intravitreal Aflibercept injection

INTERVENTIONS:
Drug: Intravitreal Aflibercept injection — Six number of injections at baseline, 1M, 2M, 3M, 4M, and 5M
  Other Names: Eylea

SUMMARY:
Retinal nonperfusion drives vision-threatening complications such as pathological neovascularization, which can lead to neovascular glaucoma, vitreous hemorrhage, or tractional retinal detachments and macular edema in diabetic retinopathy. Thus, decreasing nonperfusion area with aid of anti-VEGF agents might be a useful way to prevent deteriorating course of diabetic retinopathy. The main purpose of this study is to determine the efficacy of intravitreal aflibercept injection in improvement of retinal nonperfusion and identify associated factors in patients with nonproliferative diabetic retinopathy with moderate retinal nonperfusion.

DETAILED DESCRIPTION:
Retinal nonperfusion drives vision-threatening complications such as pathological neovascularization, which can lead to neovascular glaucoma, vitreous hemorrhage, or tractional retinal detachments and macular edema in various retinal vascular diseases including diabetic retinopathy and retinal vein occlusion. Silva et al revealed that retinal nonperfusion area was correlated highly with diabetic retinopathy severity in their recent paper. It should be clarified that retinal nonperfusion is not synonymous with retinal ischemia, which implies tissue hypoxia, but is a useful surrogate.

Retinal nonperfusion has known to be associated with the production of vascular endothelial factor (VEGF). Recently, Campochiaro et al reported that neutralization of VEGF using ranibizumab improved macular edema and reversed the worsening of retinal nonperfusion in patients with retinal vein occlusion and diabetic macular edema. The precise mechanism for improved perfusion in the VEGF treated eye is uncertain. The authors suggested that VEGF exacerbates retinal ischemia by increasing leukostasis, and intravitreal anti-VEGF agents may break the feedback loop, allowing reperfusion to occur. There might be a portion of circulation that is closed but not permanently, and this reversible closure is modulated by VEGF.

The study by Campochiaro et al, however, was limited in that they reviewed retinal nonperfusion within a template consisting of the Early Treatment Diabetic Retinopathy subfields mainly confined to posterior pole of the fundus. Wide-field retinal imaging is an imaging technique that allows a view of almost 200° of the fundus in a single image. It has been well shown that wide-field scans allow the detection of peripheral pathology that may be missed on 75 degrees of achieved by montaging the Early Treatment Diabetic Retinopathy Study 7-standard fields.

To investigators knowledge, there has been no previous study evaluating the longitudinal change of retinal nonperfusion after aflibercept treatment in a larger area of the retina by taking advantage of the 200° field of view in diabetic retinopathy. The main purpose of this study is to determine the efficacy of intravitreal aflibercept injection in improvement of retinal nonperfusion and identify associated factors in patients with nonproliferative diabetic retinopathy with moderate retinal nonperfusion.

ELIGIBILITY:
Inclusion Criteria:

* A subject must meet the following criteria to be eligible for inclusion in the study:

  1. Adults ≥ 18 years with type 1 or 2 diabetes mellitus
  2. Patients diagnosed as nonproliferative diabetic retinopathy with retinal nonperfusion (Ischemic index >20%) Severe nonproliferative diabetic retinopathy - Early proliferative diabetic retinopathy
  3. Willing and able to comply with clinic visits and study-related procedures
  4. Provide a signed informed consent form

Exclusion Criteria:

* A subject who meets any of the following criteria will be excluded from the study.

  1. Systemic exclusion criteria 1. Renal failure requiring hemodialysis or peritoneal dialysis within 6 months prior to baseline or anticipated need for hemodialysis, peritoneal dialysis at any time during the study 2. Acute cardiovascular events (acute myocardiac infarction and/or cerebral infarction) within 1 year before Visit 1 3. Blood HbA1c level greater than 12% at Visit 0
  2. Ocular exclusion criteria

  <!-- -->

  1. Diabetic macular edema involving the center of the macula (Defined as the area of the center subfield of OCT, Heidelberg Spectralis: ≥305 in women; ≥320 in men) in the study eye
  2. Presence of rubeosis (neovascularization of the iris or the angle) in the study eye
  3. Any current or history of retinal diseases that affects visual acuity in the study eye
  4. Previous treatment of panretinal photocoagulation
  5. Previous treatment with anti-VEGF in study eye within 6 months before Visit 1
  6. Previous treatment with intraocular or periocular corticosteroids in the study eye within 6 months before Visit 1
  7. Previous history of intraocular surgery other than cataract surgery in the study eye
  8. Cataract surgery within 3 months before Visit 1 in the study eye
  9. Yttrium-aluminium-garnet (YAG) capsulotomy in the study eye within 1 month before Visit 1
  10. Aphakia in the study eye
  11. Elevated intraocular pressure (≥ 22 mmHg) in spite of using topical IOP lowering agents at Visit 1 or a diagnosis of glaucoma (Visual field defect corresponding to glaucomatous optic neuropathy) in the study eye
  12. Presence of a visually significant cataract in the study eye
  13. BCVA score < 34 letters in the fellow eye
  14. Hypersensitivity to aflibercept
  15. Ocular or periocular infection
  16. Active intraocular inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Improvement of retinal nonperfusion | 1 year
  Mean changes (%) of retinal nonperfusion (Ischemic index) from baseline

SECONDARY OUTCOMES:
progression of diabetic retinopathy to proliferative diabetic retinopathy (PDR) | 1 year
  Number of patients who receive rescue treatment due to PDR and time to rescue treatment due to PDR
development of diabetic macular edema | 1 year
  Number of patients who receive rescue treatment due to DME and time to rescue treatment due to DME
Factors associated with the progression of retinal nonperfusion 1 (Functional) | 1 year
  - Visual acuity parameters: Mean changes of BCVA from baseline at every 3 month visit The proportion of subjects with gaining / losing ≥ 15letters or more in BCVA
Factors associated with the progression of retinal nonperfusion 2 (Anatomical) | 1 year
  - Optical coherence tomography (OCT) parameters: Mean changes of Central Retinal Thickness (CRT) from baseline at every 3 month visit Mean changes of Central Retinal Volume from baseline at every 3 month visit Mean change subfoveal choroidal thickness (SFChT) from baseline at every 3 month visit
Factors associated with the progression of retinal nonperfusion 3 (Anatomical) | 1year
  - Fluorescein angiography (FA) parameters: Baselinenonperfusion area(Ischemic index) at posterior and peripheral retina Baseline degree of vascular leakage at posterior and peripheral retina

OTHER OUTCOMES:
Safety outcome; Adverse effect of intravitreal aflibercept (Eylea) injection | 1 year
  Ocular and systemic adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Young Hee Yoon, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Silva PS, Dela Cruz AJ, Ledesma MG, van Hemert J, Radwan A, Cavallerano JD, Aiello LM, Sun JK, Aiello LP. Diabetic Retinopathy Severity and Peripheral Lesions Are Associated with Nonperfusion on Ultrawide Field Angiography. Ophthalmology. 2015 Dec;122(12):2465-72. doi: 10.1016/j.ophtha.2015.07.034. Epub 2015 Sep 6. PMID 26350546
- [Background] Campochiaro PA, Wykoff CC, Shapiro H, Rubio RG, Ehrlich JS. Neutralization of vascular endothelial growth factor slows progression of retinal nonperfusion in patients with diabetic macular edema. Ophthalmology. 2014 Sep;121(9):1783-9. doi: 10.1016/j.ophtha.2014.03.021. Epub 2014 Apr 24. PMID 24768239
- [Background] Silva PS, Cavallerano JD, Haddad NM, Kwak H, Dyer KH, Omar AF, Shikari H, Aiello LM, Sun JK, Aiello LP. Peripheral Lesions Identified on Ultrawide Field Imaging Predict Increased Risk of Diabetic Retinopathy Progression over 4 Years. Ophthalmology. 2015 May;122(5):949-56. doi: 10.1016/j.ophtha.2015.01.008. Epub 2015 Feb 19. PMID 25704318
- [Derived] Kim YJ, Yeo JH, Son G, Kang H, Sung YS, Lee JY, Kim JG, Yoon YH. Efficacy of intravitreal AFlibercept injection For Improvement of retinal Nonperfusion In diabeTic retinopathY (AFFINITY study). BMJ Open Diabetes Res Care. 2020 Oct;8(1):e001616. doi: 10.1136/bmjdrc-2020-001616. PMID 33077475